CLINICAL TRIAL: NCT00961623
Title: Characterizing Knee Pain and Response to Surgery Using Local Biomarkers
Status: Withdrawn | Type: Observational
Why Stopped: funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jason L. Dragoo, Principle Investigator, Stanford University
Other Study IDs: SU-07292009-3441; IRB 16305 (Other: Stanford IRB)
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial fluid lavage.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The diagnosis and monitoring of clinically-significant pathologies of the knee remains challenging, and it is unknown why only some injuries become painful or respond to surgical intervention. The limitations of diagnostic magnetic resonance imaging result in arthroscopy that is not always beneficial. Elucidation of biochemical pathways underlying pain in this condition may aid patient selection for surgery and provide pharmacotherapeutic targets. Cytokines or a novel yet uncharacterized protein may be involved in pain following meniscus injury and diagnostic cytokine assay may help physicians differentiate patients that may benefit from arthroscopy from those that may not. Additionally, evaluating post-operative biochemical profiles may provide a method of monitoring surgical outcome and understanding post-operative continuation or remission of pain.

DETAILED DESCRIPTION:
Lavage of the operative and contralateral knee for comparison are performed under anesthesia prior to arthroscopy by the infusion of 10cc sterile saline into the knee joint followed by the immediate withdrawal into the syringe, and storage at -80°C in a tube containing a protease inhibitor. At 12wk post-operative a 10cc lavage is performed on the knee that underwent surgery. Clinical findings for each sample are quantified using gold-standard symptom severity questionnaires.

The specimens will be analyzed for 31 potential biomarkers using a multiplexed immunoassay panel, the results of which will be compared with pre- and post-operative clinical findings and radiographic imaging. Plans do not currently include microarray analysis, but this may be later included.

ELIGIBILITY:
Inclusion Criteria:

•Adult patients with knee pain (acute or chronic) who had failed conservative treatment and elected for arthroscopic management. Indications for surgery included the presence of mechanical symptoms on history, a physical examination positive for McMurray's maneuver or joint line tenderness or both, absence of severe joint space narrowing on plain radiography, and the presence of grade III signal changes on MRI in an anatomic location consistent with the history and physical examination.

Exclusion Criteria:

* Less than 18 years old.
* Recent (within three months) intra-articular corticosteroid injection and past or current medical history of autoimmune disease (i.e. rheumatoid arthritis).
* In addition, no patients involved in a worker's compensation claim or personal injury litigation were enrolled in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population includes adult males and females presenting to a single orthopaedic surgeon for arthroscopic management of acute or chronic knee pain due to a mechanical derangement discernable by MRI.
  Subjects are selected using a probability sampling scheme, such that every knee arthroscopy patient that presents, without exclusionary criteria described above, is offered enrollment in the study. To date, approximately 85% of patients consent to enrollment, with no apparent sampling bias. Additionally, we are using repeated measures (matched random sampling) to evaluate the role of mediators of knee pain, and to assess the potential of utilizing expression profiles to monitor surgical outcome. For example, clinical indicators and biomarker expression profiles taken peri-operatively are compared to those obtained 12 weeks post-operatively in the same subject.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Surgical outcome: pain and functionality | 12-24wk post-operative.

SECONDARY OUTCOMES:
Expression profiles of inflammatory mediators | 24wk

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Dragoo, MD, Principal Investigator — Stanford University; Eric Leroux, Study Chair — Stanford University; Amy Wasterlain, Study Chair — Stanford University; Gaetano Scuderi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States